CLINICAL TRIAL: NCT05109702
Title: A Phase 3, Multicenter, Randomized, Double Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of Tanfanercept (HL036) Ophthalmic Solution 0.25% Compared to Placebo in Subjects With Dry Eye
Brief Title: A Study to Assess the Efficacy and Safety of Tanfanercept (HL036) Ophthalmic Solution in Participants With Dry Eye
Acronym: VELOS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL036-DED-US-P302
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Run-in (Other): Participants self-administered placebo ocular drops, twice daily (BID) in both eyes for 14 days in the Placebo Run-in Period.
  Interventions: Drug: Placebo
- 0.25% Tanfanercept Ophthalmic Solution (Experimental): Participants self-administered tanfanercept 0.25 percent (%) ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks in Treatment Period.
  Interventions: Drug: 0.25% Tanfanercept Ophthalmic Solution
- Placebo (Placebo Comparator): Participants self-administered tanfanercept placebo (vehicle solution) solution as topical ophthalmic drops, BID for up to 8 weeks in Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.25% Tanfanercept Ophthalmic Solution — Tanfanercept ophthalmic solution.
  Other Names: HL036
  Arms: 0.25% Tanfanercept Ophthalmic Solution
Drug: Placebo — Placebo vehicle solution.
  Arms: Placebo; Placebo Run-in

SUMMARY:
The objective of this study was to compare the safety and efficacy of tanfanercept ophthalmic solution 0.25% with placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have a participant-reported history of dry eye for at least 6 months prior to Visit 1
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1
* Have a best-corrected visual acuity (BCVA) of 0.7 minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit 1
* Report a score of ≥ 2 according to the Ora Calibra® ocular discomfort & 4-symptom questionnaire in at least one of the dry eye symptoms at Visits 1 and 2
* Have a Schirmer's Test score of ≤ 10 millimeter (mm) and ≥ 1 mm in at least one eye at Visits 1 and 2
* Have a corneal fluorescein staining score ≥ 2 according to the Ora Calibra® corneal and conjunctival staining scale for grading of fluorescein staining in at least 1 of the corneal regions (inferior, superior, or central) in at least 1 eye at Visits 1 and 2
* Have a conjunctival redness score ≥ 1 according to the Ora Calibra® conjunctival redness for dry eye scale in at least 1 eye at Visits 1 and 2

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months
* Have used any cyclosporine-containing drops (such as Restasis®, Cequa®), or lifitegrast ophthalmic solution (Xiidra®) within 60 days of Visit 1
* Have any previous experience using TNF inhibitor ophthalmic solutions, such Tanfanercept Ophthalmic Solution
* Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study)
* Be a woman who is pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Cornea & Cataract Consultants of Arizona, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Inc., Newport Beach, California
  - The Eye Care Institute - Butchertown Clinical Trials, Louisville, Kentucky
  - Andover Eye Associates: Raynham, Raynham, Massachusetts
  - Center For Sight, Henderson, Nevada
  - Oculus Research, Inc., Garner, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Andover Eye Associates: Warwick, Warwick, Rhode Island
  - Advancing Vision Research, LLC., Smyrna, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the eligibility criteria were enrolled at sites in the United States.
Pre-assignment Details: Participants entered the 14-day Placebo Run-in Period prior to randomization and during the 14-day period, assessments were conducted to ascertain eligibility to enter the study. Those who qualified were randomized to receive investigational product (0.25% tanfanercept ophthalmic solution or placebo) in a double-masked fashion for 8 weeks in the Treatment Period.
Groups:
- Placebo Run-in: Participants self-administered placebo ocular drops. twice daily (BID) in both eyes for 14 days in the Placebo Run-in Period.
Period: Placebo Run-in Period (14 Days)
Arm/Group | Placebo Run-in | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Started | 260 | 0 | 0
Completed | 260 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period (8 Weeks)
Arm/Group | Placebo Run-in | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Started | 0 | 130 | 130
Completed | 0 | 116 | 122
Not Completed | 0 | 14 | 8
Not completed — Adverse Event | 0 | 5 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 3
Not completed — Administrative reasons | 0 | 1 | 1
Not completed — Other than specified | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all randomized participants.
Groups:
- 0.25% Tanfanercept Ophthalmic Solution: Participants self-administered tanfanercept 0.25% ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks in Treatment Period.
- Total: Total of all reporting groups
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.31) | 63.1 (11.20) | 62.7 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 90 | 182
  Male | 38 | 40 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 118 | 121 | 239
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 98 | 103 | 201
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Corneal Staining Score (CCSS) at Day 57
Description: CCSS was graded using the Ora Calibra® Corneal and Conjunctival Fluorescein Staining Scale. The Ora Calibra® Corneal and Conjunctival Staining Scale ranged 0 = None, 1 = Trace, 2 = Mild, 3 = Moderate, and 4 = Severe; lower score indicated improvement.
Time Frame: Baseline, Day 57 (Week 8)
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 130 | 130
score on a scale
  Baseline | 2.40 (0.497) | 2.37 (0.477)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.82 (0.812) | -0.79 (0.806)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; The Least Square (LS) means, LS mean difference, Standard Errors (SEs), two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the Mixed model repeated measures (MMRM) model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.764, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.214 to 0.157], Standard Error of Mean 0.094

2. Primary Outcome: Change From Baseline in Eye Dryness Score (EDS) Assessed by Visual Analogue Scale at Day 57
Description: Eye dryness score was scored on a Visual Analogue Scale (VAS) that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline, Day 57 (Week 8)
Population: ITT population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of dryness
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 130 | 130
percentage of dryness
  Baseline | 66.1 (22.95) | 60.8 (25.57)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -16.19 (30.625) | -19.79 (26.317)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.144, MMRM; LS Mean Difference = 4.34, 95% CI 2-sided [-1.483 to 10.155], Standard Error of Mean 2.969

3. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Central Region
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of fluorescein staining. The score ranged from 0 to 4 (0=none and 4=severe), and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.43 (0.649) | -0.59 (0.667)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.45 (0.814) | -0.61 (0.723)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.57 (0.788) | -0.64 (0.861)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.82 (0.812) | -0.79 (0.806)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Week 1 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.056, MMRM; LS Mean Difference = 0.18, 95% CI 2-sided [-0.005 to 0.363], Standard Error of Mean 0.094
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Week 2 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.064, MMRM; LS Mean Difference = 0.17, 95% CI 2-sided [-0.010 to 0.359], Standard Error of Mean 0.094
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Week 4 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.328, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.093 to 0.279], Standard Error of Mean 0.095
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Week 8 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.837, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.208 to 0.168], Standard Error of Mean 0.096

4. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Superior Region
Description: as for outcome 3
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.21 (0.572) | -0.20 (0.639)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.22 (0.805) | -0.21 (0.705)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.25 (0.731) | -0.25 (0.753)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.37 (0.747) | -0.33 (0.729)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.686, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.123 to 0.187], Standard Error of Mean 0.079
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.680, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.123 to 0.188], Standard Error of Mean 0.079
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.529, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.107 to 0.207], Standard Error of Mean 0.080
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.745, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.132 to 0.185], Standard Error of Mean 0.081

5. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Inferior Region
Description: as for outcome 3
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.14 (0.611) | -0.13 (0.684)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.10 (0.732) | -0.24 (0.729)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.12 (0.756) | -0.15 (0.770)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.33 (0.708) | -0.27 (0.892)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.765, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.141 to 0.192], Standard Error of Mean 0.085
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.053, MMRM; LS Mean Difference = 0.16, 95% CI 2-sided [-0.002 to 0.331], Standard Error of Mean 0.085
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.552, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.117 to 0.219], Standard Error of Mean 0.086
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.593, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.216 to 0.124], Standard Error of Mean 0.087

6. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Temporal Region
Description: as for outcome 3
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.16 (0.742) | -0.13 (0.749)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.14 (0.870) | -0.19 (0.785)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.17 (0.875) | -0.27 (0.756)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.20 (0.746) | -0.40 (0.827)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.884, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.183 to 0.158], Standard Error of Mean 0.087
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.474, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.109 to 0.233], Standard Error of Mean 0.087
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.202, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.060 to 0.285], Standard Error of Mean 0.088
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.013, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [0.047 to 0.396], Standard Error of Mean 0.089

7. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Nasal Region
Description: as for outcome 3
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.12 (0.703) | -0.16 (0.700)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.17 (0.860) | -0.23 (0.797)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.19 (0.817) | -0.27 (0.822)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.19 (0.829) | -0.33 (0.879)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.604, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.131 to 0.224], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.519, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.119 to 0.236], Standard Error of Mean 0.091
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.299, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.085 to 0.275], Standard Error of Mean 0.092
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.124, MMRM; LS Mean Difference = 0.14, 95% CI 2-sided [-0.039 to 0.324], Standard Error of Mean 0.093

8. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Corneal Sum
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of fluorescein staining. The score ranged from 0 to 4 (0=none and 4=severe), and lower score indicated improvement. Fluorescein total staining score for corneal regions was derived as the sum of the reported scores for the inferior, superior, and central regions. Total score ranged between 0 to 12, and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.78 (1.370) | -0.91 (1.585)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.76 (1.929) | -1.06 (1.750)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.94 (1.877) | -1.04 (1.976)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -1.52 (1.904) | -1.39 (2.049)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.293, MMRM; LS Mean Difference = 0.23, 95% CI 2-sided [-0.196 to 0.647], Standard Error of Mean 0.215
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.094, MMRM; LS Mean Difference = 0.36, 95% CI 2-sided [-0.062 to 0.783], Standard Error of Mean 0.215
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.404, MMRM; LS Mean Difference = 0.18, 95% CI 2-sided [-0.245 to 0.608], Standard Error of Mean 0.217
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.806, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.485 to 0.377], Standard Error of Mean 0.220

9. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Conjunctival Sum
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of fluorescein staining. The score ranged from 0 to 4 (0=none and 4=severe), and lower score indicated improvement. Fluorescein total staining score for conjunctival regions was derived the sum of the reported scores for the nasal and temporal regions. Total score ranged between 0 to 8, and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.28 (1.219) | -0.29 (1.184)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.31 (1.582) | -0.42 (1.371)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.36 (1.463) | -0.54 (1.352)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.39 (1.427) | -0.74 (1.510)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.824, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.273 to 0.343], Standard Error of Mean 0.157
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.437, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.186 to 0.431], Standard Error of Mean 0.157
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.193, MMRM; LS Mean Difference = 0.21, 95% CI 2-sided [-0.105 to 0.519], Standard Error of Mean 0.159
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.024, MMRM; LS Mean Difference = 0.36, 95% CI 2-sided [0.048 to 0.679], Standard Error of Mean 0.161

10. Secondary Outcome: Change From Baseline in Fluorescein Staining at Weeks 1, 2, 4, and 8: Total Staining
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of fluorescein staining. The score ranged from 0 to 4 (0=none and 4=severe), and lower score indicated improvement. Fluorescein total staining score for corneal and conjunctival regions was derived as the sum of the reported scores for the inferior, superior, central, temporal, and nasal regions. Total score ranged between 0 to 20, and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -1.07 (2.104) | -1.20 (2.395)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -1.07 (3.125) | -1.48 (2.672)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -1.30 (2.974) | -1.58 (2.956)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -1.92 (2.931) | -2.12 (3.234)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.430, MMRM; LS Mean Difference = 0.26, 95% CI 2-sided [-0.386 to 0.907], Standard Error of Mean 0.329
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.143, MMRM; LS Mean Difference = 0.48, 95% CI 2-sided [-0.164 to 1.132], Standard Error of Mean 0.330
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.245, MMRM; LS Mean Difference = 0.39, 95% CI 2-sided [-0.267 to 1.042], Standard Error of Mean 0.333
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.359, MMRM; LS Mean Difference = 0.31, 95% CI 2-sided [-0.352 to 0.970], Standard Error of Mean 0.337

11. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Central Region
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of lissamine green staining. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | 0.01 (0.663) | -0.16 (0.672)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.13 (0.549) | -0.25 (0.579)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.24 (0.616) | -0.30 (0.624)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.29 (0.602) | -0.30 (0.628)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.016, MMRM; LS Mean Difference = 0.16, 95% CI 2-sided [0.030 to 0.292], Standard Error of Mean 0.067
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.099, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.021 to 0.242], Standard Error of Mean 0.067
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.493, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.086 to 0.179], Standard Error of Mean 0.068
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.987, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.133 to 0.135], Standard Error of Mean 0.068

12. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Superior Region
Description: as for outcome 11
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.11 (0.800) | -0.12 (0.523)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.20 (0.721) | -0.17 (0.576)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.25 (0.674) | -0.22 (0.549)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.18 (0.592) | -0.19 (0.656)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.655, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.109 to 0.173], Standard Error of Mean 0.072
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.826, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.157 to 0.125], Standard Error of Mean 0.072
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.861, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.155 to 0.130], Standard Error of Mean 0.073
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.556, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.101 to 0.187], Standard Error of Mean 0.073

13. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Inferior Region
Description: as for outcome 11
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.07 (0.789) | -0.14 (0.797)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.06 (0.766) | -0.33 (0.741)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.25 (0.606) | -0.27 (0.802)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.23 (0.700) | -0.33 (0.889)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.527, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.116 to 0.226], Standard Error of Mean 0.087
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.005, MMRM; LS Mean Difference = 0.25, 95% CI 2-sided [0.077 to 0.418], Standard Error of Mean 0.087
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Wek 4 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; Test type: Superiority; p = 0.920, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.164 to 0.181], Standard Error of Mean 0.088
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.286, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.080 to 0.269], Standard Error of Mean 0.089

14. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Temporal Region
Description: as for outcome 11
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.02 (0.875) | -0.18 (0.809)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.17 (0.924) | -0.25 (0.817)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.23 (0.822) | -0.31 (0.790)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.15 (0.817) | -0.17 (0.896)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.071, MMRM; LS Mean Difference = 0.18, 95% CI 2-sided [-0.015 to 0.369], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.384, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.107 to 0.278], Standard Error of Mean 0.098
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.391, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.109 to 0.280], Standard Error of Mean 0.099
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.802, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.171 to 0.222], Standard Error of Mean 0.100

15. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Nasal Region
Description: as for outcome 11
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.13 (0.735) | -0.10 (0.781)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.25 (0.962) | -0.35 (0.699)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.19 (0.775) | -0.24 (0.896)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.11 (0.926) | -0.31 (1.044)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.884, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.206 to 0.178], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.303, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.091 to 0.293], Standard Error of Mean 0.098
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.554, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.135 to 0.253], Standard Error of Mean 0.099
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.051, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [-0.001 to 0.391], Standard Error of Mean 0.100

16. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Corneal Sum
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of lissamine green staining. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Lissamine Green total staining score for corneal regions was derived as the sum of the reported scores for the inferior, superior, and central regions. Total score ranged between 0 to 12,and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.17 (1.622) | -0.42 (1.526)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.39 (1.395) | -0.75 (1.445)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.74 (1.334) | -0.79 (1.516)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.69 (1.344) | -0.82 (1.691)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.131, MMRM; LS Mean Difference = 0.26, 95% CI 2-sided [-0.077 to 0.591], Standard Error of Mean 0.170
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.040, MMRM; LS Mean Difference = 0.35, 95% CI 2-sided [0.016 to 0.685], Standard Error of Mean 0.171
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.767, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.287 to 0.389], Standard Error of Mean 0.172
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.410, MMRM; LS Mean Difference = 0.14, 95% CI 2-sided [-0.198 to 0.485], Standard Error of Mean 0.174

17. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Conjunctival Sum
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of lissamine green staining. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Lissamine Green total staining score for conjunctival regions was derived as the sum of the reported scores for the nasal and temporal regions. Total score ranged between 0 to 8, and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.14 (1.397) | -0.29 (1.261)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.42 (1.600) | -0.60 (1.307)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.42 (1.348) | -0.54 (1.488)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.26 (1.537) | -0.48 (1.717)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.324, MMRM; LS Mean Difference = 0.17, 95% CI 2-sided [-0.166 to 0.501], Standard Error of Mean 0.170
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.262, MMRM; LS Mean Difference = 0.19, 95% CI 2-sided [-0.143 to 0.525], Standard Error of Mean 0.170
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.391, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.190 to 0.485], Standard Error of Mean 0.172
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.192, MMRM; LS Mean Difference = 0.23, 95% CI 2-sided [-0.114 to 0.568], Standard Error of Mean 0.174

18. Secondary Outcome: Change From Baseline in Conjunctival Lissamine Green Staining at Weeks 1, 2, 4, and 8 : Total Staining
Description: The score for individual region was assessed by the Ora Calibra® corneal and conjunctival staining scale for grading of lissamine green staining. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Lissamine Green total staining score for corneal and conjunctival regions was derived as the sum of the reported scores for the inferior, superior, central, nasal, and temporal regions. Total score ranged between 0 to 20, and lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.32 (2.634) | -0.71 (2.252)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.81 (2.618) | -1.35 (2.277)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -1.16 (2.262) | -1.33 (2.507)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.95 (2.364) | -1.29 (2.912)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.140, MMRM; LS Mean Difference = 0.43, 95% CI 2-sided [-0.141 to 0.999], Standard Error of Mean 0.290
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.061, MMRM; LS Mean Difference = 0.55, 95% CI 2-sided [-0.025 to 1.117], Standard Error of Mean 0.291
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.490, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [-0.374 to 0.780], Standard Error of Mean 0.294
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.212, MMRM; LS Mean Difference = 0.37, 95% CI 2-sided [-0.212 to 0.953], Standard Error of Mean 0.297

19. Secondary Outcome: Change From Baseline in Conjunctival Redness Score at Weeks 1, 2, 4, and 8
Description: It was evaluated by the Ora Calibra® conjunctival redness scale for dry eye. The score ranged from 0 to 4 (0=none and 4=severe), where lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.10 (0.450) | -0.08 (0.519)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | -0.14 (0.435) | -0.19 (0.456)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -0.13 (0.577) | -0.22 (0.534)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.09 (0.648) | -0.32 (0.544)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.784, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.134 to 0.101], Standard Error of Mean 0.060
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.324, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.058 to 0.176], Standard Error of Mean 0.060
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.130, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.027 to 0.210], Standard Error of Mean 0.060
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.000, MMRM; LS Mean Difference = 0.23, 95% CI 2-sided [0.110 to 0.350], Standard Error of Mean 0.061

20. Secondary Outcome: Change From Baseline in Schirmer's Test Score at Weeks 2, 4, and 8
Description: The Schirmer test strip was placed in the lower temporal lid margin of each eye. Participants were instructed to close their eyes and after 5 minutes had elapsed, the length of moistened area of schirmer strip was recorded (millimeter [mm]) for each eye.
Time Frame: Baseline; Weeks 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 124 | 126
mm
  Change at Week 2 | 0.69 (5.155) | 0.31 (4.361)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | 1.24 (5.858) | 0.56 (4.972)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | 2.45 (5.913) | 0.51 (4.257)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.532, MMRM; LS Mean Difference = 0.39, 95% CI 2-sided [-0.834 to 1.613], Standard Error of Mean 0.623
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.252, MMRM; LS Mean Difference = 0.72, 95% CI 2-sided [-0.515 to 1.959], Standard Error of Mean 0.630
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.002, MMRM; LS Mean Difference = 1.98, 95% CI 2-sided [0.732 to 3.231], Standard Error of Mean 0.636

21. Secondary Outcome: Change From Baseline in Tear Film Break-up Time at Weeks 1, 2, 4, and 8
Description: Sodium fluorescein solution was instilled into each eye and participants were instructed to blinked several times. The time it took to form micelles from the time that the eye is opened was noted.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
seconds
  Change at Week 1 | 0.45 (1.643) | 0.55 (1.513)
  Change at Week 2: number analyzed (Participants) | 124 | 126
  Change at Week 2 | 0.17 (1.168) | 0.42 (1.171)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | 0.16 (1.064) | 0.57 (1.600)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | 0.52 (1.548) | 0.48 (1.226)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.723, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.386 to 0.268], Standard Error of Mean 0.167
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.254, MMRM; LS Mean Difference = -0.19, 95% CI 2-sided [-0.519 to 0.137], Standard Error of Mean 0.167
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.034, MMRM; LS Mean Difference = -0.36, 95% CI 2-sided [-0.690 to -0.028], Standard Error of Mean 0.169
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.640, MMRM; LS Mean Difference = 0.08, 95% CI 2-sided [-0.255 to 0.414], Standard Error of Mean 0.171

22. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Burning/Stinging
Description: Participants rated ocular symptom of burning/stinging by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of burining/stinging
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of burining/stinging
  Change at Week 1 | -7.49 (27.712) | -5.43 (21.630)
  Change at Week 2 | -8.74 (26.961) | -9.66 (23.478)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -11.84 (29.437) | -9.04 (22.261)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -12.17 (28.441) | -11.82 (22.174)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Test type: Superiority — Week 1 : The LS means, LS mean difference, SEs, two-sided 95% CIs, and pvalues of the LS mean difference will be reported from the MMRM model. MMRM p-value calculated using the final model defined for the primary analysis endpoints, including terms for baseline, grouped sites, visit (as categorical term), treatment group and the interaction of treatment group and visit as fixed effects with correlated errors; p = 0.615, MMRM; LS Mean Difference = 1.45, 95% CI 2-sided [-4.223 to 7.133], Standard Deviation 2.893
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.097, MMRM; LS Mean Difference = 4.81, 95% CI 2-sided [-0.866 to 10.494], Standard Deviation 2.894
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.718, MMRM; LS Mean Difference = 1.06, 95% CI 2-sided [-4.690 to 6.810], Standard Deviation 2.930
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.298, MMRM; LS Mean Difference = 3.09, 95% CI 2-sided [-2.728 to 8.903], Standard Error of Mean 2.963

23. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Foreign Body Sensation
Description: Participants rated ocular symptom of foreign body sensation by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of foreign body sensation
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of foreign body sensation
  Change at Week 1 | -4.63 (23.060) | -4.06 (23.349)
  Change at Week 2 | -7.93 (23.489) | -8.26 (22.783)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -7.83 (25.806) | -6.90 (22.919)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -7.81 (30.745) | -11.58 (25.182)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.343, MMRM; LS Mean Difference = 2.67, 95% CI 2-sided [-2.854 to 8.191], Standard Error of Mean 2.814
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.188, MMRM; LS Mean Difference = 3.71, 95% CI 2-sided [-1.813 to 9.232], Standard Error of Mean 2.814
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.371, MMRM; LS Mean Difference = 2.55, 95% CI 2-sided [-3.040 to 8.143], Standard Error of Mean 2.849
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.017, MMRM; LS Mean Difference = 6.92, 95% CI 2-sided [1.259 to 12.573], Standard Error of Mean 2.883

24. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Itching
Description: Participants rated ocular symptom of itching by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of itching
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of itching
  Change at Week 1 | -6.49 (21.885) | -5.52 (20.820)
  Change at Week 2 | -8.39 (23.746) | -9.07 (21.807)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -10.31 (23.372) | -9.78 (22.738)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -11.12 (27.650) | -14.33 (21.512)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.754, MMRM; LS Mean Difference = 0.85, 95% CI 2-sided [-4.452 to 6.147], Standard Error of Mean 2.700
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.368, MMRM; LS Mean Difference = 2.43, 95% CI 2-sided [-2.865 to 7.731], Standard Error of Mean 2.700
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.621, MMRM; LS Mean Difference = 1.35, 95% CI 2-sided [-4.014 to 6.715], Standard Error of Mean 2.734
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.087, MMRM; LS Mean Difference = 4.74, 95% CI 2-sided [-0.688 to 10.168], Standard Error of Mean 2.766

25. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Blurred Vision
Description: Participants rated ocular symptom of blurred vision by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of blurred vision
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of blurred vision
  Change at Week 1 | -5.95 (20.483) | -7.53 (18.674)
  Change at Week 2 | -8.94 (21.564) | -8.61 (22.511)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -9.50 (25.051) | -9.49 (22.681)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -9.24 (26.069) | -9.46 (23.783)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.110, MMRM; LS Mean Difference = 4.23, 95% CI 2-sided [-0.958 to 9.425], Standard Error of Mean 2.646
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.315, MMRM; LS Mean Difference = 2.66, 95% CI 2-sided [-2.535 to 7.855], Standard Error of Mean 2.647
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.318, MMRM; LS Mean Difference = 2.67, 95% CI 2-sided [-2.582 to 7.928], Standard Deviation 2.678
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.303, MMRM; LS Mean Difference = 2.79, 95% CI 2-sided [-2.525 to 8.111], Standard Error of Mean 2.710

26. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Eye Dryness
Description: Participants rated ocular symptom of eye dryness by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of eye dryness
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of eye dryness
  Change at Week 1 | -6.98 (22.840) | -9.23 (21.209)
  Change at Week 2 | -10.34 (23.308) | -12.52 (22.974)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -13.64 (26.572) | -13.12 (23.297)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -16.19 (30.625) | -19.79 (26.317)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.136, MMRM; LS Mean Difference = 4.44, 95% CI 2-sided [-1.402 to 10.273], Standard Error of Mean 2.975
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.165, MMRM; LS Mean Difference = 4.13, 95% CI 2-sided [-1.700 to 9.966], Standard Error of Mean 2.972
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.665, MMRM; LS Mean Difference = 1.30, 95% CI 2-sided [-4.600 to 7.207], Standard Error of Mean 3.008
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.099, MMRM; LS Mean Difference = 5.02, 95% CI 2-sided [-0.950 to 10.995], Standard Error of Mean 3.043

27. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Photophobia
Description: Participants rated ocular symptom of photophobia by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of photophobia
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of photophobia
  Change at Week 1 | -6.57 (22.155) | -3.56 (22.871)
  Change at Week 2 | -7.17 (22.689) | -5.54 (23.594)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -8.20 (28.014) | -9.10 (26.350)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -10.71 (30.328) | -12.18 (28.722)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.861, MMRM; LS Mean Difference = 0.51, 95% CI 2-sided [-5.232 to 6.254], Standard Error of Mean 2.926
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.548, MMRM; LS Mean Difference = 1.76, 95% CI 2-sided [-3.983 to 7.497], Standard Error of Mean 2.925
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.180, MMRM; LS Mean Difference = 3.97, 95% CI 2-sided [-1.839 to 9.777], Standard Error of Mean 2.960
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.189, MMRM; LS Mean Difference = 3.93, 95% CI 2-sided [-1.941 to 9.807], Standard Error of Mean 2.993

28. Secondary Outcome: Change From Baseline in Visual Analogue Scale at Weeks 1, 2, 4, and 8 : Pain
Description: Participants rated ocular symptom of pain by placing a vertical mark on VAS that ranged from 0%-100% (0=no discomfort; 100=maximal discomfort).
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: percentage of pain
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
percentage of pain
  Change at Week 1 | -6.27 (22.501) | -5.63 (18.611)
  Change at Week 2 | -5.00 (23.843) | -7.25 (19.041)
  Change at Week 4: number analyzed (Participants) | 121 | 124
  Change at Week 4 | -6.27 (29.718) | -8.27 (20.666)
  Change at Week 8: number analyzed (Participants) | 119 | 120
  Change at Week 8 | -7.23 (27.317) | -9.83 (22.370)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.613, MMRM; LS Mean Difference = 1.32, 95% CI 2-sided [-3.799 to 6.438], Standard Error of Mean 2.608
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.083, MMRM; LS Mean Difference = 4.53, 95% CI 2-sided [-0.586 to 9.653], Standard Error of Mean 2.609
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.165, MMRM; LS Mean Difference = 3.67, 95% CI 2-sided [-1.508 to 8.851], Standard Error of Mean 2.639
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.110, MMRM; LS Mean Difference = 4.28, 95% CI 2-sided [-0.964 to 9.522], Standard Error of Mean 2.672

29. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) at Weeks 1, 2, 4, and 8
Description: OSDI was a simple 12-question survey that rated the severity of the participant's dry eye disease based on the symptoms. Each question response ranged from 0 to 4, where 0 = None of the Time, 1 = Some of the Time, 2 = Half of the Time, 3 = Most of the Time, and 4 = All of the Time. Total OSDI score = (Sum of all answered questions) * 25/ (number of questions answered); which ranged from 0 to 100, with higher score representing greater disability.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -3.13 (13.229) | -5.65 (14.785)
  Change at Week 2 | -4.85 (16.092) | -6.23 (14.617)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -4.54 (18.002) | -8.16 (15.170)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -6.74 (18.702) | -9.99 (14.215)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.041, MMRM; LS Mean Difference = 3.57, 95% CI 2-sided [0.154 to 6.994], Standard Error of Mean 1.743
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.122, MMRM; LS Mean Difference = 2.70, 95% CI 2-sided [-0.723 to 6.118], Standard Error of Mean 1.743
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.009, MMRM; LS Mean Difference = 4.60, 95% CI 2-sided [1.146 to 8.056], Standard Error of Mean 1.760
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.024, MMRM; LS Mean Difference = 4.04, 95% CI 2-sided [0.544 to 7.536], Standard Error of Mean 1.781

30. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort Scale at Weeks 1, 2, 4, and 8
Description: It was assessed by the Ora Calibra® ocular discomfort scale. The score ranged from 0 to 4 (0=none and 4=severe), where lower score indicated improvement.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.22 (1.177) | -0.31 (1.084)
  Change at Week 2 | -0.34 (1.172) | -0.41 (1.060)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -0.48 (1.294) | -0.39 (1.110)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.53 (1.261) | -0.71 (1.083)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.282, MMRM; LS Mean Difference = 0.14, 95% CI 2-sided [-0.115 to 0.394], Standard Error of Mean 0.130
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.353, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.134 to 0.375], Standard Error of Mean 0.130
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.764, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.297 to 0.218], Standard Error of Mean 0.131
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.104, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [-0.044 to 0.476], Standard Error of Mean 0.133

31. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire at Weeks 1, 2, 4, and 8 : Burning Discomfort
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye included rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of burning at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data will be analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.44 (1.304) | -0.23 (1.409)
  Change at Week 2 | -0.42 (1.277) | -0.29 (1.338)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -0.56 (1.477) | -0.35 (1.238)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.55 (1.511) | -0.55 (1.304)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.969, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.300 to 0.288], Standard Error of Mean 0.150
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.504, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.194 to 0.394], Standard Error of Mean 0.150
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.915, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.281 to 0.314], Standard Error of Mean 0.152
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.195, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [-0.102 to 0.499], Standard Error of Mean 0.153

32. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire at Weeks 1, 2, 4, and 8 : Dryness Discomfort
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye included rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of dryness at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data will be analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.34 (1.048) | -0.34 (1.234)
  Change at Week 2 | -0.43 (1.266) | -0.43 (1.268)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -0.60 (1.334) | -0.44 (1.314)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.66 (1.446) | -0.74 (1.262)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.287, MMRM; LS Mean Difference = 0.16, 95% CI 2-sided [-0.133 to 0.449], Standard Error of Mean 0.148
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.260, MMRM; LS Mean Difference = 0.17, 95% CI 2-sided [-0.124 to 0.458], Standard Error of Mean 0.148
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.987, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.296 to 0.291], Standard Error of Mean 0.150
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.143, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [-0.075 to 0.519], Standard Error of Mean 0.151

33. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire at Weeks 1, 2, 4, and 8 : Grittiness Discomfort
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye included rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of grittiness at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data will be analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.26 (1.231) | -0.29 (1.278)
  Change at Week 2 | -0.45 (1.478) | -0.56 (1.293)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -0.48 (1.421) | -0.38 (1.214)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.58 (1.441) | -0.59 (1.302)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = -0.198, MMRM; LS Mean Difference = 0.19, 95% CI 2-sided [-0.102 to 0.490], Standard Error of Mean 0.151
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.076, MMRM; LS Mean Difference = 0.27, 95% CI 2-sided [-0.028 to 0.564], Standard Error of Mean 0.151
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.656, MMRM; LS Mean Difference = 0.07, 95% CI 2-sided [-0.231 to 0.367], Standard Error of Mean 0.152
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.324, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.150 to 0.454], Standard Error of Mean 0.154

34. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire at Weeks 1, 2, 4, and 8 : Stinging Discomfort
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye included rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of stinging at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: Baseline; Weeks 1, 2, 4, and 8
Population: ITT population with available data will be analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 125 | 126
score on a scale
  Change at Week 1 | -0.30 (1.193) | -0.31 (1.365)
  Change at Week 2 | -0.34 (1.191) | -0.52 (1.250)
  Change at Week 4: number analyzed (Participants) | 122 | 124
  Change at Week 4 | -0.50 (1.362) | -0.50 (1.370)
  Change at Week 8: number analyzed (Participants) | 119 | 121
  Change at Week 8 | -0.50 (1.371) | -0.61 (1.254)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.477, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.182 to 0.390], Standard Error of Mean 0.146
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.033, MMRM; LS Mean Difference = 0.31, 95% CI 2-sided [0.026 to 0.598], Standard Error of Mean 0.146
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.374, MMRM; LS Mean Difference = 0.13, 95% CI 2-sided [-0.158 to 0.420], Standard Error of Mean 0.147
Statistical Analysis 4: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.114, MMRM; LS Mean Difference = 0.24, 95% CI 2-sided [-0.056 to 0.529], Standard Error of Mean 0.149

35. Secondary Outcome: Ora Calibra® Drop Comfort Assessment at Week 1
Description: Ora Calibra® drop comfort scale ranged from 0 to 10. A score of 0 indicated comfortable and 10 indicated uncomfortable. Lower score indicated better comfort level. Immediately Upon Instillation, 1 Minute Post Instillation and 2 Minutes Post Instillation at Week 1
Time Frame: Week 1
Population: ITT population with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% Tanfanercept Ophthalmic Solution | Placebo
Number analyzed (Participants) | 124 | 126
score on a scale
  Immediately Upon Instillation at Week 1 | 2.55 (2.673) | 2.72 (2.532)
  1 Minute Post Instillation at Week 1 | 1.95 (2.063) | 2.21 (2.174)
  2 Minutes Post Instillation at Week 1 | 1.56 (1.884) | 1.79 (2.058)
Statistical Analysis 1: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; Immediately Upon Instillation at Week 1; Test type: Superiority; p = 0.598, t-test, 2 sided; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.822 to 0.475], Standard Error of Mean 0.329
Statistical Analysis 2: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; 1 Minute Post Instillation at Week 1; Test type: Superiority; p = 0.343, t-test, 2 sided; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.783 to 0.273], Standard Error of Mean 0.268
Statistical Analysis 3: Comparison: 0.25% Tanfanercept Ophthalmic Solution vs Placebo; 2 Minutes Post Instillation at Week 1; Test type: Superiority; p = 0.359, t-test, 2 sided; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.721 to 0.262], Standard Error of Mean 0.250

ADVERSE EVENTS:
Time Frame: Placebo Run-in arm: From enrollment up to Day 14 of Placebo Run-in Period 0.25% Tanfanercept Ophthalmic Solution arm and Placebo arm: From first dose up to Week 8 of Treatment Period
Description: Placebo Run-in arm: All the enrolled participants were included.
  0.25% Tanfanercept Ophthalmic Solution arm and Placebo arm: Safety population included all randomized participants who received at least one dose of the investigational product.
  Placebo Run-in arm reports all AEs; 0.25% Tanfanercept Ophthalmic Solution arm and Placebo arm reports TEAEs.
  Treatment emergent AEs (any event that occurred or worsened on or after the day the randomized study treatment was initiated) were reported.
Groups:
- Placebo Run-in: Participants self-administered placebo ocular drops BID in both eyes for 14 days in the Placebo Run-in Period.
Arm/Group | Placebo Run-in | 0.25% Tanfanercept Ophthalmic Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/260 | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/130 | 1/130
Other Adverse Events (participants affected / at risk) | 7/260 | 42/130 | 39/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Run-in (N=260) | 0.25% Tanfanercept Ophthalmic Solution (N=130) | Placebo (N=130)
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Run-in (N=260) | 0.25% Tanfanercept Ophthalmic Solution (N=130) | Placebo (N=130)
Visual acuity reduced (Eye disorders) | 0 | 10 | 9
Conjunctivitis allergic (Eye disorders) | 0 | 5 | 0
Eye discharge (Eye disorders) | 0 | 2 | 1
Vision blurred (Eye disorders) | 0 | 2 | 1
Vitreous detachment (Eye disorders) | 0 | 2 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Eyelid haematoma (Eye disorders) | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Instillation site pain (General disorders) | 0 | 14 | 15
Instillation site lacrimation (General disorders) | 0 | 1 | 0
Instillation site pruritus (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Follicular lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05109702/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT05109702/SAP_001.pdf